CLINICAL TRIAL: NCT06502834
Title: Effect of 4 Weeks of Oral D. Piger on Safety, Pharmacokinetics and Ethanol Metabolism in Overweight Individuals (2023)
Acronym: PIGER
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Max Nieuwdorp (Other)
Responsible Party: Sponsor-Investigator, Max Nieuwdorp, Principal Investigator, Amsterdam University Medical Center (UMC), Location Academic Medical Center (AMC)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023.0787
Record Dates: First submitted 2024-05-20; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Metabolic Syndrome; Steatosis of Liver
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Fatty Liver

STUDY DESIGN:
Intervention Model Description: 2x10 participants will be randomly allocated to placebo or d piger suspension once daily.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The pharmacist will provide the study intervention to the investigator in a coded fashion. Both the investigator and the participant are blinded.
  In case of emergency, an unblinding protocol is activated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo vial (10ml of glycerol 10% and 10% maltrodextrin)
  Interventions: Dietary Supplement: Placebo
- D piger (Experimental): D. piger vial with 109 colony forming units (CFU) (=108 CFU D. piger per ml in 10ml of glycerol 10% and 10% maltrodextrin).
  Interventions: Dietary Supplement: D piger

INTERVENTIONS:
Dietary Supplement: D piger — Probiotic d piger
  Arms: D piger
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of the study is to determine the effect of supplementation of the d piger strain on intestinal ethanol production in individuals with overweight.

The investigators will perform a randomized trial in 2x10 participants to measure effects on ethanol in blood, and perform fecal analyses.

DETAILED DESCRIPTION:
The investigators perform a randomized, placebo controlled trial in 2x10 participants.

The participants will be given placebo or d piger as an oral suspension once daily for 30 days.

At baseline and after 30 days, a fructose challenge test with fomepizole, gastroduodenoscopy and MRI liver + FibroScan will be performed. Patient will attend the clinical trial unit weekly for safety visits.

The participants will be overweight males or females age 18-70 with impaired glucose tolerance.

ELIGIBILITY:
Inclusion:

Male or (postmenopausal) females

* Increased waist circumference (>102 cm men, 88>cm women)
* Insulin resistance (HOMA>2.5)
* 18-70 years

Exclusion Criteria:

* Use of systemic medication (except for paracetamol), including antibiotics and pro-/prebiotics in the past three months or during the study period.
* A history of a cardiovascular event
* A history of cholecystectomy
* Overt untreated gastrointestinal disease or abnormal bowel habits
* Liver enzymes>2.5 fold higher than the upper limit of normal range
* Smoking
* Alcohol abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Gut engraftment | 30 days
  the number of reads of d piger in feces using q pcr
adverse events | 30 days
  the number of adverse events in both groups
Renal function | 30 days
  Number of participants with a decreased kidney function, defined as a rise in serum creatinine of >26,5 micromol/L in 48 h
Occurence of anemia | 30 days
  Number of patients with Hb < 8,5 mmol/L
Changes in leucocytes | 30 days
  Number of patients with leucocytes <4,0 or >10,5 x10E9 cells/L
Changes in thrombocytes | 30 days
  Number of patients with thrombocytes <150 x 10E9 cells/
Changes in aspartate aminotransferase (AST) | 30 days
  Number of patients with AST > 43 IU/L
Changes in alanine aminotransferase (ALT) | 30 days
  Number of patients with ALT > 45 IU/L
Changes in alkaline phosphatase (ALP) | 30 days
  Number of patients with ALP > 126 IU/L
Changes in Gamma-glutamyltransferase (GGT) | 30 days
  Number of patients with GGT > 117 IU/L
Changes in total bilirubin | 30 days
  Number of patients with total bilirubin > 24 micromol/L

SECONDARY OUTCOMES:
Fructose in peripheral blood | 30 days
  Area under the curve of fructose in peripheral blood upon ingestion of 1 gram / kg unlabeled fructose in combination with 1000mg of D-fructose-13C6
Fructose metabolites in breath | 30 days
  Area under the curve of various metabolites (e.g. ethanol) will be measured in breath samples upon ingestion of 1 gram / kg unlabeled fructose in combination with 1000mg of D-fructose-13C6
Time-in-range | 30 days
  Increase in Time-in-range (TIR,%), a parameter of continuous glucose monitoring devices, where TIR can be between 0 and 100%. A higher TIR reflects a better outcome.
Continuous glucose monitoring | 30 days
  Decrease in glucose variability (GV, %), a parameter of continuous glucose monitoring devices, where GV can be between 0 and 100%. A lower GV reflects a better outcome.
Glycemic control | 30 days
  Changes in fasting glucose (mmol/L)
Dietary intake | 30 days
  Participants are asked to fill out an online dietary questionnaire for the 3 days prior to study visit 2,3,4,5 and 7
Questionnaires | 30 days
  Changes in Gastro-intestinal Quality of Life Index (GIQLI score) (points). The minimum and maximum score are 31 and 155 points respectively, and a higher score reflects a better outcome.
Intestinal microbiota composition | 30 days
  Changes from baseline of relative abundance (%) of bacterial phyla, genera and species between groups and within participants.
Fructose metabolites in feces | 30 days
  Using 24h feces, the investigators will measure fecal concentrations of fructose metabolites such as ethanol, as well as short chain fatty acids (SCFAs) and bile acids.
Fructose metabolites in urine | 30 days
  Using 24h urine, the investigators will measure fecal concentrations of fructose metabolites such as ethanol, as well as SCFAs and bile acids.
Bioreactor analyses | 30 days
  Using specific anaerobic culturing, ethanol production of fecal samples will be assessed of bacterial strains.
MRI | 30 days
  Liver fat measured by proton density fat fraction (PDFF) MRI liver
FibroScan | 30 days
  Liver stiffness measured by FibroScan

CONTACTS AND LOCATIONS:
Overall Officials: Max Nieuwdorp, prof dr, Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Amsterdam UMC location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No